CLINICAL TRIAL: NCT03064737
Title: Bacterial and Human Biomarkers of Prognostic Value for Severe Legionnaire's Disease
Acronym: Proglegio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0131
Record Dates: First submitted 2016-09-02; First posted 2017-02-27 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Legionella

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This study is a non-drug one arm study (Other): Skin biopsy for genetic analyze
  Interventions: Other: Skin biopsy for genetic analyze

INTERVENTIONS:
Other: Skin biopsy for genetic analyze — It will be offered to a subgroup of adult patients carrying genetic markers predisposing to the severity of the LD infection, a skin biopsy in order to realize genetic analyses.
  This visit will be conducted once the results of genetic markers obtained (between 30 and 36 months), a specific consent will be required to patients.
  The skin biopsy will be performed according to the Clinical Department use.

SUMMARY:
Legionnaires' disease (LD) is a relatively common pneumonia in France (1200 cases/year), 98% of cases are hospitalized and 40% require intensive care unit (ICU) admission. Risk factors that may predispose to acquisition of LD are well known. Some studies suggest that genetic factor may also enhance susceptibility to LD.

The mortality rate remains high (10% to 33% in ICUs) despite improved diagnostic and therapeutic management of patients. Few prospective studies have assessed the factors associated with LD outcomes, particularly death, and most of them involved a limited number of patients.

In a multicentre cohort study, the investigators recently identified risk factors associated with higher mortality such as female sex, age, ICU stay, renal failure, corticosteroid treatment and enhanced pro-inflammatory status, as assessed by higher C-reactive protein level (PMID: 22005914). Other factors are suspected but their involvement has not been formally demonstrated including a high infectious bacterial load, particular virulence of Legionella strain, and an in vivo selection of mutants resistant to prescribed antibiotics. Disease progression is highly variable from one patient to another, and usually remains unpredictable. There are no objective criteria to predict the prognosis of these patients.

The clinical course of patients with LD remains difficult to predict because no predictive biomarkers have yet been characterized and the demonstration of the presence of mutants to antibiotics in vivo has never been done.

The main objective of the study is to correlate the L. pneumophila load (detected by PCR) to the clinical outcome of the LD infection. Clinical severity will measured by the SOFA score (Sepsis -Related Organ Failure Assessment) or the PELOD score (Pediatric Logistic Organ Dysfunction).

Secondary objectives are to identify new host and bacterial biomarkers associated with poor outcome of LD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with medical and biological signs of legionnaires' disease.
* Pediatric patients regardless of age but with a minimum weight of 7.5 kg with medical and biological signs of legionnaires' disease.
* Patient and/or his/her legal representative have reviewed the patient information/informed consent form and have given written informed consent.

Exclusion Criteria:

* None Legionella pneumophila Legionnaires' disease.
* Patients for whom respiratory secretions can't be obtained.
* Cases diagnosed only by serology.
* Outpatients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-08-23 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Legionnaire's disease severity measured by SOFA/PELOD score | At Hospital Output, on average 1 Day
  No other specific timeframe could be provided, it will depend on patients' condition. The study will evaluate correlation between the L. pneumophila load (quantify by molecular method) to the clinical outcome of the LD infection
Bacterial load measured by PCR | At Hospital Output, on average 1 Day
  No other specific timeframe could be provided, it will depend on patients' condition. The study will evaluate correlation between the L. pneumophila load (quantify by molecular method) to the clinical outcome of the LD infection

SECONDARY OUTCOMES:
Specific cytokine profile | Up to Day 5
  Cytokine profile will be measured at local level (pulmonary) and/ or systemic level (serum) and associated with severity
Genomic analyzes | At inclusion, up to 48 hours
  Genomic analyzes of bacterial genes will be associated with the legionella severity
Pulmonary microbiota | At inclusion, up to 48 hours
  Metagenomic approaches and NGS will be used to associate a specific microbiota, or changes in the severity of LD infection

CONTACTS AND LOCATIONS:
Overall Officials: Gérard LINA, Study Chair — Hospices Civils of Lyon
Locations (18):
- France (18):
  - CHU Amiens, Amiens
  - CHU d'Angouleme, Angoulême
  - CHRU Besancon, Besançon
  - CHU Brest, Brest
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - Hopital Edouard Heriot, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - CHU de Nantes, Nantes
  - Hôpital Saint Louis - APHP, Paris
  - Hôpital Tenon, Paris
  - APHP Hôpital Bichat, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Rennes, Rennes
  - CHU Saint Etienne, Saint-Etienne
  - CHU Strasbourg Nouvel Hôpital Civil, Strasbourg
  - CH Gustave Dron, Tourcoing